CLINICAL TRIAL: NCT06122272
Title: An Exploratory, Randomised, Open Label, Controlled, Multicentre Clinical Trial in Hong Kong to Explore the Effect of a New Nutritional Formula on Body Composition and Other Health Outcomes in Early Life.
Brief Title: An Exploratory Trial in Hong Kong to Explore the Effect of a New Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Nutricia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NELN202110A
Record Dates: First submitted 2023-06-28; First posted 2023-11-08 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test products: (Experimental): New formula for healthy term infants
  Interventions: Other: Test Formula
- Control products (Active Comparator): Standard, commercially available infant formula for healthy term infants
  Interventions: Other: Control Formula

INTERVENTIONS:
Other: Test Formula — The duration of the study for each subject from enrolment to final visit, is 12 months. Test Formula will be provided during this 12 month.
  Arms: Test products:
Other: Control Formula — The duration of the study for each subject from enrolment to final visit, is 12 months. Control Formula will be provided during this 12 month.
  Arms: Control products

SUMMARY:
This is an exploratory study with the aim to gain insight and potentially generate hypotheses on health benefits of feeding with study product. This study explores in healthy subjects the effect of feeding with the test product compared to the control product in early life.

DETAILED DESCRIPTION:
* Key exploratory objective is to find an effect on body composition.
* Other exploratory objectives are to find an effect on growth parameters.
* Safety and tolerance and the user experience will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, singleton, term born infants.
* Infants aged 6 months(± 2 weeks) at enrolment.
* Infants fed with formula (with or without additional weaning foods or drinks) before enrolment.
* Written informed consent (IC) from parent(s) and/or legally acceptable representative(s) aged ≥18 years at enrolment.

Exclusion Criteria:

* Infants who require a special diet other than Formula with intact cow's milk protein.
* Infants known or suspected to have cow's milk, fish protein, and/or soy allergy and/or lactose intolerance.
* Infants with current or previous illnesses/conditions and/or known or suspected congenital diseases or malformations which could interfere with the study outcomes, as per investigator's clinical judgement.
* Infants with previous, current, or intended participation in any other clinical study involving investigational or marketed products.
* Incapability of infants' parents and/or legally acceptable representative(s) to comply with study protocol as per the judgement of the investigator or investigator's uncertainty about the willingness or ability of parents legally acceptable representative(s) to comply with the protocol requirements.
* Employees and/or infants/family members or relatives of employees of Danone Nutricia, the participating sites, or any other nutrition company that develops Infant, Follow On or Young Child formulae.

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Body composition | Every 6 months, up to 12 months
  Fat mass (kg)

OTHER OUTCOMES:
Weight | Every 6 months, up to 12 months
  weight, unit: kg
Length | Every 6 months, up to 12 months
  length, unit: cm
BMI | Every 6 months, up to 12 months
  BMI = weight/length2, unit: kg/cm2
Product intake | Every 6 months, up to 12 months
  Study product intake: number of bottles and amount consumed per bottle

CONTACTS AND LOCATIONS:
Locations (2):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China
- Hong Kong Center for Clinical Research, Hong Kong, Hong Kong